CLINICAL TRIAL: NCT00942721
Title: Web-Based Cognitive Behavioral Intervention for Women With Postpartum Depression
Brief Title: Cognitive Behavioral Therapy Delivered Over the Internet for Women With Postpartum Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01MH084931 (NIH); R01MH084931 (NIH); 1R01MH084931-01A1 (NIH); DSIR 83-ATP
Record Dates: First submitted 2009-07-20; First posted 2009-07-21 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Postpartum Depression
Keywords: Web-based Intervention; CBT Treatment
MeSH Terms: conditions — Depression, Postpartum | interventions — Tuberculin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Web-based CBT for PPD (Experimental): Participants will receive Web-based CBT for PPD.
  Interventions: Behavioral: Web-based CBT for PPD

INTERVENTIONS:
Behavioral: Web-based CBT for PPD — A cognitive behavioral intervention that will provide participants with the following: online interactive tools to clarify their attitudes and reasons for wanting to change, information about some of the symptoms and mechanisms associated with feeling depressed during the postpartum period, and guidance on using behavioral and cognitive strategies proven to help reduce depressive symptoms

SUMMARY:
This study will develop and test a Web-based program to treat women with postpartum depression.

DETAILED DESCRIPTION:
After a woman gives birth, she will often feel anxious, depressed, or upset. For most women, these feelings go away within a week of giving birth, but for some, postpartum depression (PPD) can develop. PPD involves long-term, more severe feelings of anxiety, depression, and despair that impair normal functioning. Untreated PPD threatens both the mental health of mothers and the development of their infants, but many cases go untreated. This may be because of the stigma of mental health treatment, limited availability of programs, cost of treatment, or difficulty finding the time to schedule trips out of the home. Treatment through a Web-based program addresses all these concerns by providing a private, cost-efficient program available anywhere with computer access. This study will develop and test a Web-based version of cognitive behavioral therapy (CBT) to treat women with PPD to determine its feasibility and acceptability.

Participation in this study will last 3 months. All participants will be offered a Web-based version of CBT for PPD. The CBT program will include guided behavioral strategies for dealing with depression, online videos of women who have used these strategies, Web forums in which participants can ask questions of peers and experts, and periodic phone coaching. The program will last 6 weeks. All participants will complete assessments at baseline, post-treatment, and 3-month follow-up. Safety monitoring questionnaires will also be completed at Weeks 2 and 4 of treatment. Assessments will include clinical interviews and questionnaires related to the following: health; depression; demographics; maternal skills, stress, and self-efficacy; Internet use, experience, and self-efficacy; behavioral self-efficacy; and program acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Within 6 months postpartum
* Home access to the Internet
* Use of personal e-mail
* Score from 12 to 20, inclusive, on the Edinburgh Postnatal Depression Scale
* Diagnosed as having postpartum depression

Exclusion Criteria:

* Current diagnosis of substance abuse, bipolar disorder, or psychotic depression
* Currently receiving treatment for depressive symptoms, including antidepressant medication or psychotherapy
* Currently has suicidal intentionality, lethality, access to means, and history of suicide attempts

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Acceptability and feasibility of the Web-based treatment program for women with postpartum depression | Measured 3 and 6 months postpartum
Clinical utility of the program in ameliorating postpartum depression symptoms | Measured 3 and 6 months postpartum

SECONDARY OUTCOMES:
Women's characteristics that moderate the impact of the program | Measured 3 and 6 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Brian G. Danaher, PhD, Principal Investigator — Oregon Research Institute; Jeannette Milgrom, PhD, Principal Investigator — University of Melbourne; Scott Stuart, MD, Principal Investigator — University of Iowa
Locations (3):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Oregon Research Institute, Eugene, Oregon
- University of Melbourne, Heidelberg Heights, Victoria, Australia

REFERENCES:
- [Background] Danaher BG, Milgrom J, Seeley JR, Stuart S, Schembri C, Tyler MS, Ericksen J, Lester W, Gemmill AW, Lewinsohn P. Web-Based Intervention for Postpartum Depression: Formative Research and Design of the MomMoodBooster Program. JMIR Res Protoc. 2012 Nov 22;1(2):e18. doi: 10.2196/resprot.2329. PMID 23612274
- [Result] Danaher BG, Milgrom J, Seeley JR, Stuart S, Schembri C, Tyler MS, Ericksen J, Lester W, Gemmill AW, Kosty DB, Lewinsohn P. MomMoodBooster web-based intervention for postpartum depression: feasibility trial results. J Med Internet Res. 2013 Nov 4;15(11):e242. doi: 10.2196/jmir.2876. PMID 24191345